CLINICAL TRIAL: NCT07159659
Title: Post-operative Medium Chain Triglyceride Diet May Reduce Hospital Stay Following Lung Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Calvin Sze Hang Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCT Study Protocol version 1.1
Record Dates: First submitted 2025-08-22; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Neoplasms
Keywords: Medium Chain Triglyceride Diet; Lung Resection; Video-assisted thoracoscopic surgery
MeSH Terms: conditions — Thoracic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Patients in the control group will receive a standard hospital diet consistent with routine postoperative nutritional care after lobectomy with lymph node dissection. This diet does not include medium-chain triglyceride (MCT) supplementation and serves as a comparator to evaluate the effects of the MCT diet on postoperative recovery
- MCT diet during hospital stay (Experimental): Patients will receive a medium-chain triglyceride (MCT)-enriched diet during their hospital stay following lobectomy with lymph node dissection. The MCT diet is administered as part of the postoperative nutritional regimen to evaluate its impact on recovery outcomes
  Interventions: Dietary Supplement: MCT Diet
- MCT diet during hospital stay and 2 weeks after discharge (Experimental): Participants will receive a medium-chain triglyceride (MCT) diet during their hospital stay and for two weeks following discharge. This aims to evaluate the effects of continued MCT dietary supplementation on postoperative recovery outcomes after lobectomy with lymph node dissection
  Interventions: Dietary Supplement: MCT Diet

INTERVENTIONS:
Dietary Supplement: MCT Diet — MCT diet for patients following lung resection
  Arms: MCT diet during hospital stay; MCT diet during hospital stay and 2 weeks after discharge

SUMMARY:
Lung resection, a critical treatment for various thoracic diseases, including lung cancer, often necessitates prolonged hospitalization due to rare but severe postoperative complications such as chyle leaks, with an occurrence of 0.25%-3%, prolonging chest drainage, and delaying recovery. Therefore, effective postoperative care is essential for optimizing outcomes, reducing complications, and expediting recovery.

Recent studies have highlighted the significant potential of medium-chain triglyceride (MCT) diets, owing to their unique absorption pathway and metabolic properties. MCT contains mainly medium-chain fatty acids (MCFA), which is absorbed in the intestine and transported to the liver via the portal system instead of the lymphatic system. This helps to bypass the lymphatic system, thereby reducing the volume of lymph. MCFAs also provide better energy utilization in stressed condition since it does not require carnitine shuttle upon metabolism, which is beneficial to post-operation recovery.

Several studies have demonstrated the benefits of MCT diets in managing chyle leaks and supporting gastrointestinal recovery, particularly in conditions that strain the lymphatic system. For instance, short-term MCT-enriched diets have been associated with improved post-operation recovery of gastrointestinal, hepatic and renal functions, reduced total chest drainage volumes, and shorter hospital stay when compared to regular diet groups.

Patients with post-operative chyle leak following thoracic surgery are often given an MCT diet to reduce chest drain volume and hence shorten hospital stay. Based on the successful use of MCT diet on patients with chyle leak after lobectomy, it is hypothesized that patients with chylothorax provided with post-operative MCT diet can also shorten hospital stay by decreasing chest drainage. Therefore, a prospective and randomized trial is designed to investigate how post-operative MCT diet in lung resection patients without chylothorax may affect hospital stay and post-operative recovery.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized trial designed to investigate how a post-operative diet enriched with MCT affects recovery in patients undergoing video-assisted thoracic surgery (VATS). Medical students from the Chinese University of Hong Kong, under the supervision of the principal investigator, will conduct the study, including obtaining consent and collecting data. Experienced surgeons at the Prince of Wales Hospital will perform the VATS procedures.

2.2 Hypotheses

1. MCT diet can speed up post-operative recovery and shorten hospital length of stay.
2. MCT diet poses no adverse effects in post-operative recovery for patients without chyle leak following lung surgery.
3. The use of MCT diet after discharge for 2 weeks can enhance patient recovery and possibly reduce readmissions or complications.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria for All procedures:

1. Age between 18 - 80 years
2. Body mass index <35 kg/m2
3. Suitable for minimally invasive surgery
4. Willingness to participate as demonstrated by giving informed consent

Project-specific Criteria:

1. Patients performed lobectomy with lymph node dissection

Exclusion Criteria:

Patient general exclusion criteria:

1. Contraindication to general anesthesia
2. Severe concomitant illness that drastically shortens life expectancy or increases the risk of therapeutic intervention
3. Untreated active infection
4. Non-correctable coagulopathy
5. Emergency surgery
6. Vulnerable population (e.g. mentally disabled, pregnancy)

Project-specific Criteria

1. Segmentectomy
2. Pleurodesis
3. Esophageal procedures
4. Redo/readmitted patients for lung resection
5. Chylothorax (Triglyceride > 110 mL, excluded at day 1 routine lab check)
6. Air leak (> 30 mL/min when back to ward)
7. Heart Failure
8. Renal failure (estimated GFR < 30; CKD grading stage 4-5)
9. Moderate to severe adhesion (defined at randomization by surgeon; criteria include estimated surface area of adhesion and staging)
10. History of tuberculosis or empyema

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
hospital length of stay (LOS) | From the end of the lung resection procedure until the time of patient discharge, assessed up to 7 days post-surgery
  hospital length of stay (LOS), which is hypothesized to be reduced following the administration of an MCT diet. Currently, patients undergoing lobectomy using VATS have a median LOS of approximately 3-4 days. The study aims to investigate whether MCT diet interventions can reduce this to 2 days, representing a 30% reduction in hospital stay.

SECONDARY OUTCOMES:
Total Chest Drain Output (mL) | From the end of the lung resection procedure until the time of chest drain removal assessed up to 7 days post-surgery
  Chest drain output indirectly reflects recovery status. The total chest drain output will be measured using the Medela digital chest drainage system, which is routinely used for patients undergoing lobectomy. Compared to manual drainage system, this system allows more precise monitoring of fluid output. This information will help evaluate the overall impact of the MCT diet on postoperative recovery, particularly in reducing fluid drainage.
Patient Satisfaction and Tolerability | Upon discharge (assessed up to 7 days post-surgery), 2 weeks post discharge, 3 months post discharge
  Patient-reported outcomes will be assessed using a quality of life (QoL) questionnaire, which is an established tool for evaluating recovery after surgery. The questionnaire will include:
  * Patient satisfaction with their recovery process
  * Tolerability of the MCT diet
  * Any challenges experienced during the diet, including adherence and acceptability
Number of Participants with Symptoms Associated with MCT Diet | Upon discharge (assessed up to 7 days post-surgery), 2 weeks post discharge, 3 months post discharge
  Patients will be monitored for any gastrointestinal discomfort associated with the MCT diet, including:
  * Diarrhea
  * Constipation
  * Bloating
  * Increased flatus
  Reports of these symptoms will be collected during the hospital stay and follow-up visits to assess the safety and tolerability of the MCT diet.
Number of patients with Infection symptoms | Upon discharge (assessed up to 7 days post-surgery), 2 weeks post discharge, 3 months post discharge
  · Observing for symptoms such as fever or shortness of breath (SOB), which will be incorporated into the QoL questionnaire
Number of patients with infection risk | Upon discharge (assessed up to 7 days post-surgery), 2 weeks post discharge, 3 months post discharge
  Regular checks for pleural-based complications, such as effusion, through chest X-rays (performed before discharge and during follow-ups)

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No